CLINICAL TRIAL: NCT05145166
Title: Safety Observation of Live Attenuated Mumps Vaccines in Junior High School Students Under 14 Years Old Vaccinated With Live Attenuated Mumps Vaccines in Shanxi Province
Brief Title: Safety Study of Live Attenuated Mumps Vaccines in Junior High School Students Under 14 Years Old
Status: Completed | Type: Observational
Sponsor: Sinovac (Dalian) Vaccine Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-MUMPS-4007
Record Dates: First submitted 2021-11-25; First posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Mumps
MeSH Terms: conditions — Mumps

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — This study did not involve sample collection.Only adverse reactions/events at 30 minutes, 14 days and 30 days after vaccination of live attenuated mumps vaccine were collected by face-to-face or telephone follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Safety group — All of the participants(N=10000) received one dose of live attenuated mumps vaccine.Vaccine will given by single intramuscular injection(0.5 ml) on day 0.

SUMMARY:
This study of live attenuated mumps vaccines is an observational study in which active monitoring and passive monitoring were combined to conduct safety observation.The live attenuated mumps vaccines manufactured by Sinovac (Dalian) Vaccine Technology Co., Ltd.The purpose of this study is to evaluate the safety of live attenuated mumps vaccines after large-scale application and accumulate safety data for the application of live attenuated mumps vaccines,and provide scientific basis for the formulation of vaccine immunization prevention strategies.

DETAILED DESCRIPTION:
This study of live attenuated mumps vaccines is an observational study in which active monitoring and passive monitoring were combined to conduct safety observation.The live attenuated mumps vaccines manufactured by Sinovac (Dalian) Vaccine Technology Co., Ltd.Bao'ji, Xian'yang, Yan 'an and Han'zhong of Shaanxi Province were selected as the research center.A total of 10000 junior high school students under 14 years old who voluntarily received a dose of live attenuated mumps vaccines were be enrolled.Adverse reactions/events at 30 minutes, 14 days and 30 days after vaccination of live attenuated mumps vaccine were were collected by face-to-face or telephone follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Junior high school students under 14 years old;
* The subjects and guardians of the subjects can understand and voluntarily sign the informed consent form ;
* Subjects and their legal guardians are able to attend follow-up visits and follow all study procedures (such as cooperating in completing safety observation notes)

Exclusion Criteria:

-

Max Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: In this study, only junior high school students under 14 years old who were judged by vaccination doctors to be eligible for vaccination and voluntarily received one dose of live attenuated mumps vaccine were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
Safety index-the incidence of local and systemic adverse reactions | From 0 day to 14 days after vaccination
  The incidence of local and systemic adverse reactions from 0 day to 14 days after vaccination.
Safety index-The incidence of local and systemic adverse reactions | From 0 day to 30 days after vaccination.
  The incidence of local and systemic adverse reactions from 0 day to 30 days after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Weijun Hu, Master, Principal Investigator — Shaanxi Provincial Center for Disease Control and Prevention
Locations (3):
- China (3):
  - Baoji Center for Disease Prevention and Control, Baoji, Shanxi
  - Xianyang Center for Disease Control and Prevention, Xianyang, Shanxi
  - Yanan Center for Disease Prevention and Control, Yan’an, Shanxi

REFERENCES:
- [Derived] Hu W, Jia N, Meng W, Zhou T, Wang R, Xiong Y, Luan C, Zhang S. Safety analysis of a live attenuated mumps vaccine in healthy adolescents in China: A phase 4, observational, open-label trial. PLoS One. 2023 Sep 21;18(9):e0291730. doi: 10.1371/journal.pone.0291730. eCollection 2023. PMID 37733724